CLINICAL TRIAL: NCT03055845
Title: A Prospective, Randomised, Double-blinded, Placebo-controlled, Single Ascending Dose Study Investigating the Safety and Local Tolerability of STA363 Compared to Placebo in 15 Patients With Chronic Discogenic Low Back Pain
Brief Title: A Single Ascending Dose Study of Safety and Tolerability of STA363 Compared to Placebo in 15 Patients With Chronic Discogenic Low Back Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stayble Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STA-01; 2015-004812-39 (EudraCT Number)
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Following treatment of 2 patients in each dose group (injections with active drug and placebo, respectively), safety data will be reviewed. If no safety or tolerability concerns are identified, the next 3 patients in each dose group will be treated (active treatment or placebo [2:1]).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- STA363 dose 1 (Experimental)
  Interventions: Drug: STA363
- STA363 dose 2 (Experimental)
  Interventions: Drug: STA363
- STA363 dose 3 (Experimental)
  Interventions: Drug: STA363
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STA363 — STA363, containing 3 different doses of active ingredient, in a volume of 1.5 mL. Administered as intradiscal injection.
  Arms: STA363 dose 1; STA363 dose 2; STA363 dose 3
Drug: Placebo — Matching placebo solution with identical appearance to the test product, used as reference treatment. Administered as intradiscal injection.
  Arms: Placebo

SUMMARY:
A phase I, randomized, double-blinded, placebo-controlled, single ascending dose study to investigate the safety, local tolerability and transformation of nucleus pulposus following intradiscal injection of STA363 or placebo in patients with discogenic low back pain.

15 patients will participate in either of 3 dose groups, each comprising 5 patients:

* Group 1: STA363 dose 1 (3 patients) or placebo (2 patients)
* Group 2: STA363 dose 2 (3 patients) or placebo (2 patients)
* Group 3: STA363 dose 3 (3 patients) or placebo (2 patients)

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-related procedures
* Chronic discogenic low back pain present for more than 6 months prior to the screening visit
* 20 to 60 years of age at the screening visit
* Insufficient response to at least 6 months of non-operative treatment (analgesics and/or antiinflammatory medication, physiotherapy etc.)
* A single lumbar disc appropriate for treatment at L3/4 to L5/S1, based on clinical evaluation by the investigator
* Pfirrmann grade II-III
* Ability to understand the written and verbal information about the study

Exclusion Criteria:

* Treatment with any investigational product within 3 months prior to the screening visit
* More than one painful intervertebral disc
* A painful intervertebral disc above L3/4 level
* Current infection or prior history of spinal infection (e.g., discitis, septic arthritis, epidural abscess) or an active systemic infection
* Previous lumbar spine surgery
* Previous disc invasive treatment procedures at the affected level(s) (e.g., intradiscal electrothermal therapy, intradiscal radiofrequency thermocoagulation)
* Pfirrmann grade I, IV and V
* Evidence of prior lumbar vertebral body fracture or trauma
* Need for spinal decompression assessed by the investigator
* Presence of disc extrusion or sequestration
* Patients previously included in the study
* Patients suffering from psychosomatic pain in the opinion of the investigator
* Referred leg pain of compressive origin
* Known alcohol and/or drug abuse
* Severe intercurrent illness (e.g. rheumatic disease or chronic pain syndrome) or concomitant treatment (e.g. immunosuppressive drugs), which, in the opinion of the investigator, may put the patient at risk when participating in the study, or affect the patient's ability to take part in the study
* Clinically significant abnormalities in clinical chemistry or haematology parameters as assessed by the investigator
* Pregnant or lactating females or intention to become pregnant within the study period
* Known allergy to any of the components of the drug product or placebo
* Known opioid allergy or intolerance
* Patients requiring treatment with warfarin or other anticoagulant therapy
* Unwillingness to refrain from treatment with non-steroidal anti-inflammatory drugs (NSAIDs) within 5 days before the planned study treatment
* Body weight less than 50 kg

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Local injection site reactions | Up to 4 weeks after injection
Frequency and severity of adverse events | Up to 12 weeks after injection
Changes in routine safety laboratory parameters | Up to 12 weeks after injection
Visual analogue scale (VAS) pain (injection site) | Up to 15 minutes after injection
Changes in vital signs | Up to 12 weeks after injection
Changes in electrocardiogram (ECG) | 1 day after injection
Changes in physical examination findings | 1 and 12 weeks after injection
Changes in body weight | 12 weeks after injection

SECONDARY OUTCOMES:
Transformation of nucleus pulposus into connective tissue by magnetic resonance imaging (MRI) | 12 weeks after injection
Disc height by MRI | 12 weeks after injection

OTHER OUTCOMES:
VAS pain (leg and back) | 1, 4 and 12 weeks after injection
Oswestry disability index (ODI) score | 12 weeks after injection

CONTACTS AND LOCATIONS:
Locations (1):
- Stockholm Spine Center, Löwenströmska Sjukhuset, Upplands Vasby, Sweden